CLINICAL TRIAL: NCT04908085
Title: Creating Satisfying Engagement in Daily Life Through Coaching for People With Multiple
Brief Title: Creating Satisfying Engagement in Daily Life Through Coaching for People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dorothy Kessler (Other)
Responsible Party: Sponsor-Investigator, Dorothy Kessler, Assistant Professor, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 6032454
Record Dates: First submitted 2021-05-19; First posted 2021-06-01 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis; Quality of Life
Keywords: Coaching
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Waitlist control trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPC (Experimental): Occupational Performance Coaching delivered by telephone
  Interventions: Behavioral: Occupational Performance Coaching
- Waitlist control (No Intervention): Intervention provided after post intervention assessment

INTERVENTIONS:
Behavioral: Occupational Performance Coaching — Six sessions of OPC delivered by telephone over 10 weeks.
  Other Names: OPC
  Arms: OPC

SUMMARY:
Multiple sclerosis (MS) is a complex disease that negatively impacts a person's ability to participate in a wide range of important and meaningful activities1-4. MS rehabilitation interventions often focus on reducing symptoms, with the assumption that fewer symptoms will lead to improved participation in daily activities5-8. Yet, literature shows that engagement in necessary and desired activities requires more than symptom reduction - it requires people with chronic diseases like MS to apply their knowledge and skills to a complex self-management process9-11 that balances personal values, and activity and environmental demands. Core self-management skills include self-monitoring, problem-solving, decision-making, goal setting, action planning, and the ability to adjust plans when necessary12. Looking beyond MS, coaching interventions have enabled people with stroke13-16, traumatic brain injury17, and Parkinson's disease18, 19 to develop self-management skills and achieve personally meaningful activity goals. Occupational Performance Coaching (OPC) is a well-developed form of coaching that builds competence in core self-management skills and improves participation in daily activities20, 21. The investigator's preliminary work indicates that OPC is an acceptable and feasible intervention for people with MS22. The investigators now must determine if OPC reduces the impact of MS on participation in daily activities and increases the satisfaction of people with MS in performance of personally important daily activities. Therefore, the investigators will conduct a waitlist-control randomized clinical trial (RCT) with 30 adults with MS to determine if receipt of six OPC sessions improves participants' satisfaction with performance in daily activities (primary outcome). The investigators will also examine whether OPC reduces illness intrusiveness (MS impact), improves resilience, and improves autonomy and participation (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* able to participate in coaching in English.

Exclusion Criteria:

1. serious cognitive impairment as indicated by a score of 10 or more on the Short Blessed Test,
2. severe depression as measured by the PHQ-2
3. are receiving life, health or executive coaching by a certified coach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure | Pre-intervention, 10 weeks, and 2 months post intervention
  Measure of performance and satisfaction with performance and satisfaction on a scale of 1-10 where 10 indicates higher performance or satisfaction with performance.

SECONDARY OUTCOMES:
Illness Intrusiveness Rating Scale | Pre-intervention, 10 weeks, and 2 months post intervention
  The Illness Intrusiveness Rating Scale captures induced interference of chronic disease and treatment on valued activities and interests. The scale is a brief self-report questionnaire that is composed of 13 items: health, diet, work, active recreation, passive recreation, financial situation, relationship with your spouse, sex life, family relations, other social relations, self-expression/ self-improvement, religious expression, and community and civic involvement. Respondents rate the degree to which their illness and/or treatment interfere with these domains using a seven-point scale (1- not very much, 7 - very much). A higher overall score (range13-91) indicates a higher level of illness intrusiveness.
MS Impact Scale-29 | Pre-intervention, 10 weeks, and 2 months post intervention
  The MS Impact scale is a 29-item scale that measures the impact of MS on day-to day life on a scale from 1 (not at all) to 5 (extremely). Higher scores (range 29-145) indicate higher impact of MS on daily life.
Connor-Davidson Resilience Scale-10 | Pre-intervention, 10 weeks, and 2 months post intervention
  The CDRS is a 10 item questionnaire used to measure participant's perception of their ability to cope and adapt to challenges. Scores range from 0-40 where a higher score indicates better resilience.
Impact on Participation and Autonomy Questionnaire | Pre-intervention, 10 weeks, and 2 months post intervention
  The IPA provides a measure of limitations in participation and autonomy. The tool includes 39 questions across 5 domains: autonomy indoors, autonomy outdoors, family role, social life and relationships, and work and education. Participants rate each item on scale from 0 (very good) to 4 (very poor). Score range is 0-156 with higher scores representing poorer autonomy and participation.

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Kessler, Principal Investigator — Queen's University
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kessler D, Franz M, Malakouti N, Rajachandrakumar R, Baharnoori M, Finlayson M. Randomized Controlled Trial of Occupational Performance Coaching for Adults With Multiple Sclerosis. Arch Phys Med Rehabil. 2024 Sep;105(9):1649-1656. doi: 10.1016/j.apmr.2024.05.022. Epub 2024 Jun 6. PMID 38851554